CLINICAL TRIAL: NCT01814280
Title: Differentiated Intervention Aimed at Reducing Medication Errors on Basis of an Individual Risk Assessment - a Pilot Study
Brief Title: Reducing Medication Errors on Basis of an Individual Risk Assessment
Acronym: MERIS1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MERIS1
Record Dates: First submitted 2012-08-16; First posted 2013-03-19 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Drug Safety
Keywords: Medication errors; Medication review; Risk stratification; Patient safety
MeSH Terms: interventions — Medication Review

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Medication review (Other): Medication review performed by either a clinical pharmacist or a clinical pharmacologist
  Interventions: Other: Medication review

INTERVENTIONS:
Other: Medication review — Medication review performed by either a clinical pharmacist or a clinical pharmacologist

SUMMARY:
Background:

Medication reviews performed on admission to hospitals reduce medication errors; however, evidence of effect on morbidity and mortality is currently inconsistent. It is known that patients' risks of experiencing medication errors are dependent on both patient- and drug factors, e.g. age, co-morbidity, number of drugs, risk of side effects.

Aim and hypothesis:

The aim of this pilot study is to study acute medical patients' risk of getting a medication error based on an algorithm that takes into account both patient and drug related factors. Secondary, the investigators will explore whether our methods are applicable in a randomised controlled trial. The investigators will also decide the number of patients in a randomised controlled trial based on this pilot study.

The hypothesis is that an algorithm that has already been developed can stratify patients according to their risk of experiencing a medication error.

Methods:

100 acute admitted patients will be risk stratified at admission (>8 hours after). The patients who have highest risks of medication errors will receive a medication review performed by either a clinical pharmacist or a clinical pharmacologist.

ELIGIBILITY:
Inclusion Criteria:

* Acutely admitted patients
* Age>17 years

Exclusion Criteria:

* Dying patients
* Suicial patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Medication errors | During the patients' hospital stay
  The patients' electronic medical record will be assessed for medication errors during the patients' hospitalization. It will be assesed by a clinical pharmacologist to assess the validity of the algorithm. Medication errors are defined as errors in prescriptions that either harm or have the potential to harm the patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital,, Aarhus, Denmark